CLINICAL TRIAL: NCT02545205
Title: New Technology for Individualised, Intensive Training of Gait After Stroke- Phase II Trials, Study I
Brief Title: New Technology for Individualised, Intensive Training of Gait After Stroke Study I
Acronym: HAL-RCT-II
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Stopped due to limited access to medical technology devices.
Sponsor: Danderyd Hospital (Other)
Collaborators: University of Tsukuba (Other); Sahlgrenska University Hospital (Other); Umeå University (Other)
Responsible Party: Principal Investigator, Susanne Palmcrantz, PhD, Reg. Physiotherapist, Danderyd Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HAL-RCT-Phase II-Study I
Record Dates: First submitted 2015-08-24; First posted 2015-09-09 (Estimated); Last update posted 2023-02-13 (Actual); Status verified 2018-04

CONDITIONS: Stroke; Ambulation Difficulty; Hemiparesis
Keywords: Rehabilitation; Robotics
MeSH Terms: conditions — Stroke; Mobility Limitation; Paresis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hybrid Assistive Limb (HAL) (Experimental)
  Interventions: Device: Hybrid Assistive Limb (HAL)
- Conventional gait training (Active Comparator)
  Interventions: Other: Conventional gait training

INTERVENTIONS:
Device: Hybrid Assistive Limb (HAL) — Intensive gait training with Hybrid Assistive Limb (HAL) is performed, 1 session/day, 4 days/week during 4 weeks. Time for each session is individualised but does not exceed 60 minutes/session (effective walking time with HAL).
  Arms: Hybrid Assistive Limb (HAL)
Other: Conventional gait training — The conventional gait training is performed according to current best evidence based practice and may include over ground walking with assistance and/or assistant devices as well as the use of a treadmill and body weight support and training of gait function in activities of daily living.
  Arms: Conventional gait training

SUMMARY:
The overall purpose of this project is to establish the added value of training with the Hybrid Assistive Limb (HAL) exoskeleton system as part of regular rehabilitation intervention programs after stroke.

The aim of this study is to explore if HAL training when combined with conventional training in the subacute stage after stroke may accelerate the recovery of independence in walking when compared to conventional training only and if recovery is related to stroke lateralization?

DETAILED DESCRIPTION:
Patients will be randomized using a block randomization by a nurse, who is not otherwise involved in the study, into either 1) HAL training in addition to the conventional program or 2) evidence based conventional gait training only. The block randomization will be designed so that an even number of patients with left and right sided hemiparesis will have been included in each group at the end of the study.

Conventional training (including gait practice) will be performed according to current best practice (approximately 30-60 min per day, 5 days per week) and may include stepping, weight shifting, over ground walking as well as the use of a treadmill with/without body weight support (BWS).

HAL training will be performed 4 days a week for 4 weeks (i.e. 16 sessions) with the single-leg version of HAL, primarily by use of the voluntary HAL-mode (CVC mode), on a treadmill with BWS. The therapist(s) educated in the HAL method will optimize the HAL settings for each individual during each session, in order to obtain a symmetrical gait pattern as close to normal gait as possible.

Outcomes The primary outcome will be changes in the FAC-score during the intervention. FAC assesses activity in terms of independence in walking on a six-grade-ordinal-scale ranging from non-functional walking to independent walking outside. During the intervention assessments with the FAC will be performed weekly by the patients' physiotherapist responsible for conventional rehabilitation. This therapist will otherwise not be involved in the study.

Secondary outcomes include aspects of body functions assessed by use of the NIH Stroke Scale, Albert's test, Fugl-Meyer Assessment(FMA-LE) and the Modified Ashworth Scale for the lower extremities.

Activities and Participation will be assessed by use of Functional Ambulation Categories, 2 minutes walk test in self-preferred speed, Berg Balance Scale, Barthel Index and EQ5D.

Patients' perception of training will be assessed by a study specific questionnaire.

Adverse events (such as irritated skin, pain, falls) will be documented continuously in the study protocol according to a specific study form.

Assessments will be performed 1) before and 2) after the intervention with 3) a follow up at 6 months.

ELIGIBILITY:
Patients aged 18-67 will be recruited from 1) the University Department of Rehabilitation Medicine at Danderyd Hospital in Stockholm and 2) Sahlgrenska University Hospital in Gothenburg, where they are admitted to inpatient rehabilitation early after stroke. Inclusion criteria will be: less than 8 weeks since stroke onset; inability to walk independently due to lower extremity paresis (i.e. Functional Ambulation Categories (FAC) score 0-1), able to sit on a bench with or-without supervision at least 5 minutes; sufficient postural control to allow upright position in standing with aids and/or manual support; ability to understand training instructions as well as written and oral study information and to express informed consent; body size compatible with the HAL suit. Exclusion criteria include: contracture restricting gait movements at any lower limb joint; cardiovascular or other somatic condition incompatible with intensive gait training; and severe, contagious infections.

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Change in Functional Ambulation Categories (FAC) | Assessed at baseline, weekly, after 4 weeks of intervention and at 6 months post intervention
  Level of independence in walking, range 0-5

SECONDARY OUTCOMES:
Objectively quantify the impairment caused by a stroke, using the National Institutes of Health Stroke Scale (NIHSS) | At baseline
Fugl-Meyer for Lower extremities | Assessed at baseline, after 4 weeks of intervention and at 6 months post intervention
  Sensory and motor function in lower extremities
Albert's test | Assessed at baseline
  Spatial negelct
2 Minutes Walk Test (MWT) | Assessed at baseline, after 4 weeks of intervention and at 6 months post intervention
  Walking
Berg Balance scale | Assessed at baseline, after 4 weeks of intervention and at 6 months post intervention
  Balance
Barthel Index | Assessed at baseline, after 4 weeks of intervention and at 6 months post intervention
  Independence in mobility and personal care
Perception of the intervention | after 4 weeks of intervention
  Interview, Study group using Hybrid Assistive Limb (HAL) only.
Stroke Impact Scale (SIS) | Assessed at 6 months after intervention
  Functioning and disability, Interview
EQ-5D | Assessed at baseline, after 4 weeks of intervention and at 6 months post intervention
  Health Outcome

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Department of Rehabilitation Medicine, Danderyd Hospital, Danderyd, Stockholm County
  - Sahlgrenska University Hospital, Gothenburg

REFERENCES:
- [Background] Nilsson A, Vreede KS, Haglund V, Kawamoto H, Sankai Y, Borg J. Gait training early after stroke with a new exoskeleton--the hybrid assistive limb: a study of safety and feasibility. J Neuroeng Rehabil. 2014 Jun 2;11:92. doi: 10.1186/1743-0003-11-92. PMID 24890413
- [Background] Wall A, Borg J, Palmcrantz S. Clinical application of the Hybrid Assistive Limb (HAL) for gait training-a systematic review. Front Syst Neurosci. 2015 Mar 25;9:48. doi: 10.3389/fnsys.2015.00048. eCollection 2015. PMID 25859191